CLINICAL TRIAL: NCT03936400
Title: Development of Therapeutic Conversations With Females Diagnosed With Cancer and Their Partners: Evaluation of Effectiveness in Adjustment of Sexuality and Intimacy
Brief Title: Development of Therapeutic Conversations With Females Diagnosed With Cancer and Their Partners
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erla Kolbrún Svavarsdóttir (Other)
Collaborators: Landspitali University Hospital (Other)
Responsible Party: Sponsor-Investigator, Erla Kolbrún Svavarsdóttir, Professor, University of Iceland
Organization: University of Iceland (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UIceland-22019JIJ
Record Dates: First submitted 2019-04-10; First posted 2019-05-03 (Actual); Last update posted 2019-11-22 (Actual); Status verified 2019-11

CONDITIONS: Cancer
Keywords: cancer; females; partners
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Randomized controlled trial (Experimental): Experimental group receiving a couple-based intervention
  Interventions: Behavioral: Couple-based intervention and and evaluation of effectiveness in increasing adjustment of sexuality and intimacy
- Active comparator: control group (Active Comparator): A control group that receives same but delayed couple-based intervention
  Interventions: Behavioral: Couple-based intervention and and evaluation of effectiveness in increasing adjustment of sexuality and intimacy

INTERVENTIONS:
Behavioral: Couple-based intervention and and evaluation of effectiveness in increasing adjustment of sexuality and intimacy — Three face-to-face therapeutic conversations and an optional web-based evidence based information (about sexual consequences of cancer treatment)

SUMMARY:
The main purpose of the doctoral study is to better understand the experience of cancer diagnosis and treatment in how it effects sexuality and intimacy of the female cancer patient and her partner.

DETAILED DESCRIPTION:
With this increased understanding, an intervention, comprised of therapeutic interventions with the couple, will be conducted and assessed on how it affects the couple's general well-being and recovery of the sexual and intimate relationship.

The intervention consists of three therapeutic conversations, based on the Illness Beliefs model in family nursing, and an optional web-based evidence based information. The aim of the intervention is to support the facilitating beliefs of the couple in adapting to changes in intimacy and identify constraining beliefs. In the first session an emphasis is on creating an optimal context for changing beliefs by building good therapeutic relationship and to invite them to share their experience, giving them the opportunity to voice their own concerns and reflect on how their situation effects their intimate relationship. In the second session, the couple take a closer look at what they themselves deem important in adjusting to changes in their intimate relationship. In both sessions information about the possible sexual side effects of treatment will be offered as needed and evidence based, optional web-based information on practical solutions will be provided. In the booster-session, the couple will assess how they have been adjusting in their intimate relationship and any positive changes that have occurred will be accentuated.

ELIGIBILITY:
Inclusion Criteria:

* All females, 18 yrs and older, diagnosed with cancer (all types) and their partners
* Have began cancer treatment (surgical treatment, chemotherapy, radiation) - Are in a couple relationship
* Live in Iceland and are able to travel to site of intervention
* Speak and write Icelandic

Exclusion Criteria:

* Single females
* Do not read or write nor speak Icelandic

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Females (hetrosexual, homosexual) and their partners.
Enrollment: 120 (Actual)
Dates: Start 2017-04-15 (Actual); Primary Completion 2019-08-20 (Actual); Study Completion 2019-08-20 (Actual)

PRIMARY OUTCOMES:
Sexual Concerns Questionnaire-Gynecological Cancer (SCQ-GC) at baseline in experimental group (T1). | T1 ( at baseline).
  This questionnaire is a survivor self-report that screens for sexual concerns after cancer.
Sexual Concerns Questionnaire-Gynecological Cancer (SCQ-GC) post-intervention in experimental group (T2). | T2 (1-2 weeks after baseline).
  This questionnaire is a survivor self-report that screens for sexual concerns after cancer.
Sexual Concerns Questionnaire-Gynecological Cancer (SCQ-GC) post-intervention in experimental group (T3). | T3 (3 months after baseline).
  This questionnaire is a survivor self-report that screens for sexual concerns after cancer.
Sexual Concerns Questionnaire-Gynecological Cancer (SCQ-GC) at baseline in control group (T1). | T1 (at baseline).
  This questionnaire is a survivor self-report that screens for sexual concerns after cancer.
Sexual Concerns Questionnaire-Gynecological Cancer (SCQ-GC) pre-intervention in control group (T2). | T2 (wait-pre-intervention, 1 month after baseline).
  This questionnaire is a survivor self-report that screens for sexual concerns after cancer.
Sexual Concerns Questionnaire-Gynecological Cancer (SCQ-GC) post-intervention in control group (T3). | T3 (post-intervention, 1-2 weeks from T2).
  This questionnaire is a survivor self-report that screens for sexual concerns after cancer.
Sexual Concerns Questionnaire-Gynecological Cancer (SCQ-GC) post-intervention in control group (T4). | T4 (post-intervention, 3 months from T3).
  This questionnaire is a survivor self-report that screens for sexual concerns after cancer.
Partnership Questionnaire (PFB; Partnerschaftsfragebogen) at baseline in experimental group (T1). | T1 (at baseline).
  This 30-item questionnaire was developed for diagnosis and evaluation in conjoint marital therapy.
Partnership Questionnaire (PFB; Partnerschaftsfragebogen) post-intervention in experimental group (T2). | T2 (1-2 weeks after baseline).
  This 30-item questionnaire was developed for diagnosis and evaluation in conjoint marital therapy.
Partnership Questionnaire (PFB; Partnerschaftsfragebogen) post-intervention in experimental group (T3). | T3 (3 months after baseline).
  This 30-item questionnaire was developed for diagnosis and evaluation in conjoint marital therapy.
Partnership Questionnaire (PFB; Partnerschaftsfragebogen) at baseline in control group (T1). | T1 (at baseline).
  This 30-item questionnaire was developed for diagnosis and evaluation in conjoint marital therapy.
Partnership Questionnaire (PFB; Partnerschaftsfragebogen) pre-intervention in control group (T2). | T2 (wait-pre-intervention, 1 month after baseline).
  This 30-item questionnaire was developed for diagnosis and evaluation in conjoint marital therapy.
Partnership Questionnaire (PFB; Partnerschaftsfragebogen) post-intervention in control group (T3). | T3 (post-intervention, 1-2 weeks from T2).
  This 30-item questionnaire was developed for diagnosis and evaluation in conjoint marital therapy.
Partnership Questionnaire (PFB; Partnerschaftsfragebogen) post-intervention in control group (T4). | T4 (post-intervention, 3 months from T3).
  This 30-item questionnaire was developed for diagnosis and evaluation in conjoint marital therapy.
ICE-Beliefs questionnaire for couples (ICE-COUPLE) at baseline in experimental group (T1). | T1 ( at baseline).
  The instrument measures changes in facilitating or constraining beliefs through Therapeutic conversation intervention (TCI).
ICE-Beliefs questionnaire for couples (ICE-COUPLE) post-intervention in experimental group (T2). | T2 (1-2 weeks after baseline).
  he instrument measures changes in facilitating or constraining beliefs through Therapeutic conversation intervention (TCI).
ICE-Beliefs questionnaire for couples (ICE-COUPLE) post-intervention in experimental group (T3). | T3 (3 months after baseline).
  The instrument measures changes in facilitating or constraining beliefs through Therapeutic conversation intervention (TCI).
ICE-Beliefs questionnaire for couples (ICE-COUPLE) at baseline in control group (T1). | T1 (at baseline).
  The instrument measures changes in facilitating or constraining beliefs through Therapeutic conversation intervention (TCI).
ICE-Beliefs questionnaire for couples (ICE-COUPLE) pre-intervention in control group (T2). | T2 (wait-pre-intervention, 1 month after baseline).
  The instrument measures changes in facilitating or constraining beliefs through Therapeutic conversation intervention (TCI).
ICE-Beliefs questionnaire for couples (ICE-COUPLE) post-intervention in control group (T3). | T3 (post-intervention, 1-2 weeks from T2).
  The instrument measures changes in facilitating or constraining beliefs through Therapeutic conversation intervention (TCI).
ICE-Beliefs questionnaire for couples (ICE-COUPLE) post-intervention in control group (T4). | T4 (post-intervention, 3 months from T3).
  The instrument measures changes in facilitating or constraining beliefs through Therapeutic conversation intervention (TCI).
The Illness Intrusiveness Rating Scale (IIRS) at baseline in experimental group (T1). | T1 ( at baseline).
  Illness Intrusiveness Rating Scale (IIRS) measures the extent to which disease and/or its treatment interferes with lifestyles, activities and interests.
The Illness Intrusiveness Rating Scale (IIRS) post-intervention in experimental group (T2). | T2 (1-2 weeks after baseline).
  Illness Intrusiveness Rating Scale (IIRS) measures the extent to which disease and/or its treatment interferes with lifestyles, activities and interests.
The Illness Intrusiveness Rating Scale (IIRS) post-intervention in experimental group (T3). | T3 (3 months after baseline).
  Illness Intrusiveness Rating Scale (IIRS) measures the extent to which disease and/or its treatment interferes with lifestyles, activities and interests.
The Illness Intrusiveness Rating Scale (IIRS) at baseline in control group (T1). | T1 (at baseline).
  Illness Intrusiveness Rating Scale (IIRS) measures the extent to which disease and/or its treatment interferes with lifestyles, activities and interests.
The Illness Intrusiveness Rating Scale (IIRS) pre-intervention in control group (T2). | T2 (wait-pre-intervention, 1 month after baseline).
  Illness Intrusiveness Rating Scale (IIRS) measures the extent to which disease and/or its treatment interferes with lifestyles, activities and interests.
The Illness Intrusiveness Rating Scale (IIRS) post-intervention in control group (T3). | T3 (post-intervention, 1-2 weeks from T2).
  Illness Intrusiveness Rating Scale (IIRS) measures the extent to which disease and/or its treatment interferes with lifestyles, activities and interests.
The Illness Intrusiveness Rating Scale (IIRS) post-intervention in control group (T4). | T4 (post-intervention, 3 months from T3).
  Illness Intrusiveness Rating Scale (IIRS) measures the extent to which disease and/or its treatment interferes with lifestyles, activities and interests.

CONTACTS AND LOCATIONS:
Overall Officials: Ása Þórisdóttir, PhD, Study Chair — University of Iceland
Locations (1):
- University of Iceland, School of Health Sciences, Faculty of Nursing, Reykjavik, Iceland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jonsdottir JI, Vilhjalmsson R, Svavarsdottir EK. Effectiveness of a couple-based intervention on sexuality and intimacy among women in active cancer treatment: A quasi-experimental study. Eur J Oncol Nurs. 2021 Jun;52:101975. doi: 10.1016/j.ejon.2021.101975. Epub 2021 May 11. PMID 34020136
- [Derived] Jonsdottir JI, Vilhjalmsson R, Svavarsdottir EK. The Benefit of a Couple-Based Intervention Among Women in Active Cancer Treatment on Sexual Concerns: A Quasi-Experimental Study. Cancer Nurs. 2021 Nov-Dec 01;44(6):E589-E599. doi: 10.1097/NCC.0000000000000949. PMID 33899783